CLINICAL TRIAL: NCT05381961
Title: Observational Study of Bioimpedance Spectroscopy (BIS) for Use in a Renal Population
Brief Title: Observational Study of BIS in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ImpediMed Limited (Industry)
Collaborators: California Institute of Renal Research (Other); Frenova Renal Research (Other)
Responsible Party: Sponsor
Other Study IDs: IPD-ESRD-001
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Kidney Failure, Chronic; Renal Failure Chronic; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Stable hemodialysis regimen: Up to 50 patients on hemodialysis >6 months, with stable target/dry weight, and have not been hospitalized recently
  Interventions: Device: Bioimpedance spectroscopy (BIS) measurement, SOZO device
- Unstable hemodialysis regimen: Up to 20 patients who have been on hemodialysis <6 months, or have unintended weight loss/gain, or have recently been hospitalized
  Interventions: Device: Bioimpedance spectroscopy (BIS) measurement, SOZO device

INTERVENTIONS:
Device: Bioimpedance spectroscopy (BIS) measurement, SOZO device — All patients enrolled in this study will undergo BIS measurement before and after 12 hemodialysis sessions (pre-dialysis and post-dialysis BIS measurements for each session). Measurements are not provided to treating physicians and are not used to guide clinical decisions; i.e., BIS measurements are collected for observational purposes only.

SUMMARY:
This observational study will evaluate bioimpedance spectroscopy (BIS) measurements from patients undergoing hemodialysis.

DETAILED DESCRIPTION:
This observational study will evaluate bioimpedance spectroscopy (BIS) measurements from patients undergoing hemodialysis. If changes in BIS parameters correlate with changes in fluid volume and patient symptoms, BIS may help provide a non-invasive way to estimate the amount of fluid to dialyze during a hemodialysis session. Data from this study may be used to inform the design of a future interventional trial of BIS use in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years of age;
2. End-stage renal disease with a GFR <15 mL/min/1.73m^2 and dialysis dependent requiring 3-times weekly dialysis;
3. Able and willing to remove shoes and stand on SOZO for BIS measurements;
4. Able to provide written informed consent and authorization to use and disclose health information.

Exclusion Criteria:

1. Is enrolled in a concurrent interventional study of an experimental treatment that may confound the results of this study, in the investigator's opinion;
2. Has a clinical condition that would not allow them to complete the study;
3. Is pregnant or planning to become pregnant; women of childbearing potential (or premenopausal) must be on 2 forms of contraception;
4. Is lactating;
5. Has an implanted cardiac rhythm management device (pacemaker or implantable cardioverter defibrillator);
6. Has an amputation of a limb/s resulting in them being unable to make contact with the SOZO electrodes (amputations of fingers and toes are not an exclusion);
7. Patient determined by the attending physician unlikely to be compliant with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (aged 18+ years) with end-stage renal disease, are known to a study investigator, and undergo hemodialysis 3-times per week at an outpatient dialysis unit.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
BIS correlation with amount of fluid dialyzed | 12 hemodialysis sessions (over 4 to 6 weeks)
  BIS-measured fluid change (volume) will be analyzed for correlation with the volume of fluid removed during hemodialysis as documented on dialysis treatment records.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Boiskin, MD, Principal Investigator — Balboa Research
Locations (2):
- United States (2):
  - Balboa Research - Kearny Mesa, San Diego, California
  - Balboa Research - Rancho Bernardo, San Diego, California

IPD SHARING:
Plan to Share IPD: No